CLINICAL TRIAL: NCT04311489
Title: Single-center, Randomized, Double-blind, Placebo-controlled Clinical Trial for the Safety, Tolerability and Efficacy of Ularitide in Cirrhosis Patients With Refractory Ascites.
Brief Title: Refractory Ascites in Patients With Liver Cirrhosis, and the Potential Treatment With 48 Hours Infusion of Ularitide.
Acronym: ULA04
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis showing safety concerns
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); ADS AIPHIA Development Services AG (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ULA04; 2019-002268-28 (EudraCT Number)
Record Dates: First submitted 2020-03-12; First posted 2020-03-17 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2022-05

CONDITIONS: Cirrhosis, Liver; Ascites Hepatic
Keywords: Cirrhosis; Ascites; Refractory ascites; Natriuresis; Diuresis; Urodilatin; Ularitide; natriuretic peptide
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis; Ascites | interventions — Ularitide

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ularitide (Experimental): Test product. Continuous intravenous infusion with 30 ng/kg/min for 48 hours.
  Interventions: Drug: Ularitide
- Placebo (Placebo Comparator): Matching placebo. Continuous IV infusion for 48 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ularitide — Continuous intravenous infusion for 48 hours at a dose of 30 ng/kg/min. Depending on effect and/or side effects dose can be adjusted to 15 ng/kg/min or 45 ng/kg/min.
  Other Names: Urodilatin
  Arms: Ularitide
Drug: Placebo — Continuous intravenous infusion for 48 hours at a bodyweight-adjusted infusion rate.
  Arms: Placebo

SUMMARY:
This clinical trial intends to investigate the safety, tolerability and efficacy of ularitide on the renal response in patients with liver cirrhosis and refractory ascites for a maximum exposure duration of 48 hours, through a randomized, placebo-controlled, double-blind, single-center trial.

DETAILED DESCRIPTION:
The investigators hypothesize that ularitide infusion is more effective than placebo to induce and maintain clinically meaningful natriuresis and diuresis in patients with liver cirrhosis and refractory ascites.

Participants will be given ularitide or placebo intravenously while hospitalized at Department of Hepatology and Gastroenterology at Aarhus University Hospital. During the hospitalization blood and urine samples are frequently collected.

30 ng/kg/min is the starting dosage for all participants. Depending on effects and/or side effects, ULA04 is designed to individualize treatment doses by up- and/or downtitration of the infusion dose within a predefined dose range. Relevant safety precautions are incorporated in the study design and treatment will be prematurely discontinued if a pre-defined stopping criteria presents.

Patients will be followed up for the appearance of serious adverse events 30 days after the treatment.

If a separate written consent is given by the participants, additional blood and urine samples will be collected and stored in a biobank for future research.

ELIGIBILITY:
Inclusion Criteria:

* Men and women >18 years
* Liver cirrhosis confirmed by fibroscan (>20 kPa), or by imaging with signs of an irregular liver surface with collaterals, or clinically by cirrhosis stigmata
* Refractory ascites Definition: failure to respond to or intolerance to high dose diuretics (spironolactone up to 400mg/day and furosemide up to 160mg/day) and early ascites recurrence (reappearance of grade 2 or 3 ascites within 4 weeks of initial mobilization or ≥2 paracentesis within last 3 months)
* Urine sodium excretion <60 mmol/24 hour
* Serum creatinine <150 µmol/L
* Child-Turcotte-Pugh score of B or C (<13)
* Bilirubin <150 µmol/L
* Prothrombin time (PP) 0.20-0.60 (INR 1.3-2.5)
* Systolic blood pressure ≥95 mmHg
* Written informed consent to participate in the clinical trial

Exclusion Criteria:

* Gastrointestinal bleeding within 2 weeks prior to inclusion
* Proteinuria >500 mg/day
* Hemoglobin <5.5 mmol/L
* Spontaneous bacterial peritonitis within 2 weeks prior to inclusion
* Loculated ascites
* Hepatic encephalopathy grade 2-4 (West-Haven classification)
* Obstructive uropathy
* Primary kidney disease
* Known diagnosis of congestive heart failure
* Known diagnosis of acute-on-chronic liver failure
* Known diagnosis of systemic inflammatory response syndrome
* Acute infections by known diagnosis and/or antibiotic treatment
* Known HIV infection
* Known allergy to the investigational drug or other natriuretic peptides
* Treatment with dobutamine, levosimendan, milrinone, any phosphodiesterase inhibitor, octreotide, midodrine, vasopressin, dopamine or other vasopressors within 2 weeks prior to inclusion
* Nephrotoxic drugs within 1 month prior to inclusion
* Fertile women not using contraception, either an intrauterine device or hormonal contraception
* Positive pregnancy test in pre-menopausal women or in breast-feeding women
* Participation in an interventional clinical drug trial within 1 month prior to inclusion
* Legal incapacity or limited legal capacity
* Patients who are employees or relatives of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Absolute and relative change in sodium excretion rate. | After 24 hours and at termination of treatment (up to 48 hours)
Absolute and relative change in urine volume. | After 24 hours and at termination of treatment (up to 48 hours)
Change of absolute body weight. | At termination of treatment (up to 48 hours)

SECONDARY OUTCOMES:
Number of responders in the ularitide group versus the placebo group, defined by: | Throughout the treatment period. Latest measure at termination of treatment (up to 48 hours)
  Urine volume increase of ≥100 % versus baseline, urine volume increase ≥50 % versus baseline, natriuresis increase by ≥100 % versus baseline and/or body weight reduction by ≥2 kg versus baseline.
Absolute and relative change in sodium excretion rate. | After 2 hours and 4 hours of treatment and at 6 hours post-treatment follow-up
Absolute and relative change in urine volume. | After 2 hours and 4 hours of treatment and at 6 hours post-treatment follow-up
Absolute and relative change in plasma cyclic guanosine monophosphate (cGMP) concentration. | Throughout the treatment period. Latest measure at 6 hours post-treatment follow-up
Absolute and relative change in waist circumference. | After 24 hours and at termination of treatment (up to 48 hours)
Absolute and relative change in serum creatinine. | After 24 hours and at termination of treatment (up to 48 hours)
Absolute and relative change in estimated glomerular filtration rate (eGFR). | After 24 hours and at termination of treatment (up to 48 hours)
Absolute and relative change in plasma and urine osmolalities. | Throughout the treatment period. Latest measure at 6 hours post-treatment follow-up
Absolute and relative change in GFR-24h-Crea (Glomerular filtration rate based on 24-hour creatinine clearance). | After 24 hours and 48 hours of treatment
Absolute and relative change in hematocrit. | After 24 hours and 48 hours of treatment and at 6 hours post-treatment follow-up
Absolute and relative change in plasma copeptin concentration. | After 24 hours and 48 hours of treatment and at 6 hours post-treatment follow-up
Absolute and relative change in plasma renin concentration. | After 24 hours and 48 hours of treatment and at 6 hours post-treatment follow-up
Absolute and relative change in plasma angiotensin concentration. | After 24 hours and 48 hours of treatment and at 6 hours post-treatment follow-up
Absolute and relative change in plasma aldosterone concentration. | After 24 hours and 48 hours of treatment and at 6 hours post-treatment follow-up

OTHER OUTCOMES:
Incidence of adverse events/reactions. | Throughout the treatment period and until 6 hours post-treatment follow-up
Incidence of serious adverse events/reactions. | Throughout the treatment period and until 30 days post-treatment follow-up
Incidence of stopping criteria leading to a dose reduction. | Throughout the treatment period (up to 48 hours)
Incidence of stopping criteria leading to early termination of treatment. | Throughout the treatment period (up to 48 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Henning Grønbæk, Prof,MD,PhD, Principal Investigator — Department of Hepatology and Gastroenterology, Aarhus University Hospital,
Locations (1):
- Department of Hepatology and Gastroenterology, Aarhus University Hospital, Aarhus, Central Jutland, Denmark

REFERENCES:
- [Background] Carstens J, Greisen J, Jensen KT, Vilstrup H, Pedersen EB. Renal effects of a urodilatin infusion in patients with liver cirrhosis, with and without ascites. J Am Soc Nephrol. 1998 Aug;9(8):1489-98. doi: 10.1681/ASN.V981489. PMID 9697672
- [Background] Carstens J, Gronbaek H, Larsen HK, Pedersen EB, Vilstrup H. Effects of urodilatin on natriuresis in cirrhosis patients with sodium retention. BMC Gastroenterol. 2007 Jan 26;7:1. doi: 10.1186/1471-230X-7-1. PMID 17257428
- [Background] Gantzel RH, Meyer M, Mazgareanu S, Aagaard NK, Jepsen P, Holzmeister J, Watson H, Gronbaek H. Ularitide as treatment of refractory ascites in cirrhosis- a study protocol for a randomised trial. Dan Med J. 2021 Nov 12;68(12):A07210610. PMID 34851251